CLINICAL TRIAL: NCT03283228
Title: Cd11b and Cd56 as Prognostic Markers in Acute Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Z A Kamel, Dr, Assiut University
Other Study IDs: Myeloid Leukemia Markers
Record Dates: First submitted 2017-08-27; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CD11b and CD56 markers: Cd11b and Cd56 as Prognostic Markers in Acute Myeloid Leukemia
  Interventions: Diagnostic Test: Cd11b and Cd56 markers
- Haematological parameters in cases of adult AML: Study correlation between CD56 and CD11b expression with haematological parameters in cases of adult AML
  Interventions: Diagnostic Test: Cd11b and Cd56 markers

INTERVENTIONS:
Diagnostic Test: Cd11b and Cd56 markers — The expression of CD11b and CD56 in newly diadnosed cases of AML
  Other Names: Cd11b and Cd56 as Prognostic Markers in Acute Myeloid Leukemia

SUMMARY:
1. Detect the expression of marker CD56 and CD11b in newly diagnosed cases of adult AML.
2. Study correlation between CD56 and CD11b expression with haematological parameters in cases of adult AML.

DETAILED DESCRIPTION:
1. CD11b expression level is a prognostic biomarker for AML patient. CD11b positivity could predict a poor prognosis for AML patients.
2. CD56 antigen expression, an inexpensive, easy to detect and reproduce index, is closely related to the prognosis of AML patients

ELIGIBILITY:
Inclusion Criteria:

Anew diagnosis cases of adult AML

Exclusion Criteria:

1. Pediatric AML .
2. follow up cases of adult AML

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Anew diagnosis cases of adult AML
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
CD11b and CD56 marker | 24 month
  Detect the expression of marker CD56 and CD11b in newly diagnosed cases of adult AML.